CLINICAL TRIAL: NCT03435406
Title: Investigation of the Prevalence of Hepatopulmonary Syndrome in Cirrhosis Patients Caused by Hepatitis B in Western China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Lu KZ, Professor of Institute of Anesthesiology, Southwest Hospital, Third Military Medical University Affiliation: Southwest Hospital, China, Southwest Hospital, China
Other Study IDs: CEE-HBV
Record Dates: First submitted 2018-02-02; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Hepatopulmonary Syndrome
Keywords: Hepatitis B, Chronic; Cirrhosis; Hepatopulmonary Syndrome
MeSH Terms: conditions — Hepatopulmonary Syndrome; Hepatitis B, Chronic; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cirrhosis with HPS: Diagnosed as HPS
- cirrhosis without HPS: Not Diagnosed as HPS

SUMMARY:
to investigate the prevalence of hepatopulmonary syndrome in cirrhosis patients caused by Hepatitis B in western China

DETAILED DESCRIPTION:
Hepatopulmonary syndrome (HPS) occurs in approximately 4%-29% of cirrhotic patients and influences mortality. China has 100 million Hepatitis B virus (HBV) carriers and Chronic HBV infection is well-recognized risk factor for cirrhosis.But little is known about the prevalence of HPS in cirrhosis patients caused by HBV in western China. The aim of this study was to investigate the HPS incidence, and the signs, symptoms, arterial blood gas, and BMP9 in the serum of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old;
2. American association of anesthesiologists(ASA) score: I-III;
3. Ability to comply with research programmes;
4. Voluntary participation in the study;
5. Has the history of HBV infection;
6. No primary cardiopulmonary disease (heart disease, emphysema, pneumonia, asthma, etc.)

Exclusion Criteria:

1. Severe heart, lung, kidney disease coexisted;
2. American association of anesthesiologists(ASA) score≥IV; forced expiratory volume at one second (FEV1) or forced vital capacity (FVC) <70%, or FEV1 / FVC <0.70;
3. Mental state could not cooperate
4. Absence of written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were selected with cirrhosis caused by HBV including Southwest Hospital, the first affiliated hospital of Chongqing Medical University, the People's hospital of Rongchang district and Qijiang District people's hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
transthoracic contrast enhanced echocardiography (CEE) | During the operation
  through the ultrasound to evaluate the imagine of cardiac cavity after intravenous injection of agitated saline
arterial blood gas | During the operation
  arterial blood gas analysis was performed through the radial artery.
medical history | During the operation
  The medical history was collected through consultation.
acropachy | During the operation
  acropachy was examined by inspection
spider angioma | During the operation
  spider angioma was examined by inspection
liver palms | During the operation
  liver palms was examined by inspection
oxygen saturation | During the operation
  oxygen saturation was examined by pulse oximetry

SECONDARY OUTCOMES:
the content of bone morphogenetic protein (BMP9) in the patients with and without HPS | 4 to 6 months after the study completion
  the content and expression of BMP9 were determined by immunohistochemistry.
micro ribonucleic acid 144 (miR144), micro ribonucleic acid 200 (miR200) in the patients with and without HPS | 4 to 6 months after the study completion
  the content and expression of BMP9 were determined by polymerase chain reaction (PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Lu K Zhi, PhD, Study Director — Department of Anesthesiology, Southwest Hospital Third Military Medical University
Locations (1):
- Department of Anesthesiology, Southwest Hospital Third Military Medical University, Chongqing, Chongqing Municipality, China